CLINICAL TRIAL: NCT06139237
Title: Factores Que Determinan la Respuesta a la Ingesta: Efecto de la Carga Proteica
Brief Title: Factors That Determine the Responses to Food Ingestion: Protein Load
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PR(AG)338/2016P
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: meal ingestion; meal composition; postprandial responses; hedonic sensations; homeostatic sensations

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-protein supplement (Experimental): The high-protein supplements contains 47.3% protein, 39.4% carbohydrates, 13.3% lipids. A dose containing 20.8 g protein and diluted to a volume of 200 mL will be administered (187 Kcal).
  Interventions: Other: High-protein supplement
- Balanced supplement (Active Comparator): The high-protein supplements 22.2% protein, 67.85% carbohydrates, 9.95% lipids. A dose containing 20.8 g protein and diluted to a volume of 200 mL will be administered (399.3 Kcal)
  Interventions: Other: Balanced supplement

INTERVENTIONS:
Other: High-protein supplement — High protein supplement 200 mL
  Arms: High-protein supplement
Other: Balanced supplement — Balanced supplement 200 mL
  Arms: Balanced supplement

SUMMARY:
Aim: to determine to what extent meal composition influences postprandial sensations. Experimental design: randomized cross-ower study comparing the responses to a high protein (47.3% protein, 39.4% carbohydrates, 13.3% lipids) versus a balanced (22.2% protein, 67.85% carbohydrates, 9.95% lipids). In each participant the meals (both containing 20.8 g protein and diluted to a volume of 200 mL) will be tested on separate days. Healthy, non-obese participants (8 men and 8 women) will be instructed to eat a standard dinner the day before, to consume a standard breakfast at home after overnight fast, and to report to the laboratory, where the test meal will be administered 3 h after breakfast. Studies will be conducted in a quiet, isolated room with participants sitting on a chair. Perception will be measured at 5 min intervals 10 min before and 20 min after ingestion, at 10 min intervals up to 60 min after the meal and at 30 min up to 120 min after ingestion. Blood samples for biochemical and hormonal determinations will be taken before and after ingestion.

ELIGIBILITY:
Inclusion Criteria:

* non-obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in digestive well-being measured after the test meal | 1 day
  Change in average well-being measured by 10 score scales at the end of the test meal.

SECONDARY OUTCOMES:
Change in satiety measured after the test meal | 1 day
  Change in average satiety measured by 10 score scales at the end of the test meal
Change in fullness sensation measured after the test meal | 1 day
  Change in average fullness measured by 10 score scales at the end of the test meal
Change in abdominal discomfort/pain sensation measured after the test meal | 1 day
  Change in average abdominal discomfort/pain measured by 10 score scales at the end of the test meal
Change in mood measured after the test meal | 1 day
  Change in average mood measured by 10 score scales at the end of the test meal.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Spain